CLINICAL TRIAL: NCT05373329
Title: Comparison of a Mobile Digital Health Intervention Versus Waitlist Control for the Treatment of Depression and Anxiety: A Randomized Controlled Trial
Brief Title: Testing a Digital Health Intervention App for Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Sanvello (Unknown)
Responsible Party: Principal Investigator, Brenna Renn, Dr. Brenna Renn, Principal Investigator, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1691460
Record Dates: First submitted 2021-06-22; First posted 2022-05-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-guided app use (Experimental): Participants receive the self-guided app intervention immediately. All participants will have a total of 8 weeks participating in the study, and will complete assessments every 2 weeks during that 8-week period.
  Interventions: Device: Sanvello (app)
- waitlist control (No Intervention): Participants receive the self-guided intervention after an 8-week waiting period (waitlist control group). All participants will have a total of 8 weeks participating in the study, and will complete assessments every 2 weeks during that 8-week period.

INTERVENTIONS:
Device: Sanvello (app) — Sanvello is a commercially available mobile app designed to teach users strategies to manage their stress, anxiety, and depression. Users can choose which tools they want to use. The strategies are digital implementations of existing practices in psychology such as thought records, mindfulness meditation & relaxation exercises, and behavioral activation.
  Other Names: self-guided app; Sanvello Premium
  Arms: self-guided app use

SUMMARY:
Although mobile applications ("apps") for mental health are popular and widely available, little is known about how well they actually help people with common mental health symptoms of depression, anxiety, and stress. We are partnering with a commercially available app to test how well this app helps people's mental health over 8 weeks. Participants will be randomly assigned (like flipping a coin) to two groups: (a) using the app, (b) no app until after 8 weeks. We will ask participants to complete online surveys about their mood and well-being so we can better understand the effects of these different treatments.

DETAILED DESCRIPTION:
This research is focused on evaluating mental health outcomes associated with a commercially available programs offered by Sanvello Health compared to a control condition.

Background on the Sanvello program:

Sanvello is a commercially available mobile app designed to teach users strategies to manage their stress, anxiety, and depression. Users can choose which tools they want to use. The strategies are digital implementations of existing practices in psychology such as thought records, mindfulness meditation & relaxation exercises, and behavioral activation. The app also includes features like mood and health tracking to help individuals notice patterns in their moods and adjust their activities to manage their emotions more effectively. Additionally, there is a "hope board" which serves as a place for users to put inspirational quotes, reassuring photos, or save their completed activities to be reminded of their successes in using the app. Finally, the app offers a peer support community, which is a discussion board for users to connect with others going through similar experiences or who share interests. The interventions based on Cognitive-Behavioral Therapy (CBT) include the "Thoughts" tool, which educates users about the effect of thinking errors or "cognitive distortions" on emotions and then prompts users to complete a text-based thought record, identify any cognitive distortions, and then challenge those thoughts (via positive reframe). The "Goals" tool is also based on CBT and allows users to create a list of goals to face their fears (in the case of anxiety) or re-engage with life (for those struggling with depression). The tool helps users to track their tasks and progress. The interventions based on Mindfulness include "Meditations" which provides a suite of activities for users to learn mindfulness, practice deep breathing or body scans, guided relaxation activities, or simply listen to soothing sounds. Sanvello also offers health-behavior tracking which allows users to monitor activities of their choice such as caffeine consumption, exercise, time spent with loved ones, etc. Users can also track their mood state "How are you feeling?". Additionally, users can create and track custom health activities and associate words with their mood from pre-set options such as "stressed" or "happy" or can specify their own words using a hashtag such as "#engaged".

Treatment Groups:

Study participation involves assignment to one of these two groups (app use or waitlist control) and participation in study assessments. The interventions are developed, maintained, and delivered by Sanvello independent of this research study. App use is not prescribed, regulated, or restricted in any way as part of this study; rather, we are interested in collecting app use as outcome data. Primary analyses will be intent-to-treat (i.e., based on group assignment) regardless of app use; app use will also be examined as a covariate during analyses.

Although the app is commercially available, the active condition in this study (app use) require payment for regular users (i.e., those not involved in this study). We hope to incentivize participation by offering the app free to all participants, including waitlist participants (after their 8-week waiting period). Ultimately, there is no way of knowing whether a person chooses to download and use Sanvello or another commercially available digital mental health app during this trial.

Study Procedures:

This is a fully remote study. Participants in the study will be allowed to use the app however they want, in the same way that regular app users can. There is no minimum or maximum "dose" specified.

All research procedures (independent from app use) will be collected and stored in REDCap, a secure web application for building and managing online surveys and databases. This includes the consent information, screening, and assessment procedures. Participant contact data (i.e., email address) will be remotely collected and stored. They will receive a hyperlink directing to download the app once they are deemed eligible. REDCap will send reminders for each assessment timepoint with the survey link to complete the assessment. At no point is direct contact with members of the research team necessary.

Please see the uploaded image of study flow for additional visualization of these procedures ("Sanvello RCT flow"). The study procedures are as follows:

1. Online recruitment ad with link to landing page

   a. Online ads will indicate that the University of Nevada-Las Vegas and Sanvello are partnering to better understand the effectiveness of mobile apps for mental health. Recruitment from patients seeking care on the Sanvello platform will direct to a similar advertisement. Examples of the advertisements have been uploaded along with this application.
2. Basic screening and eligibility questions via online survey

   1. Verify age (18 or older)
   2. Verify US location
   3. Verify compatible smartphone use
3. Potentially eligible participants will be directed to review online consent information

   a. Participants will be asked to complete a consent quiz to ensure they understand the study protocol, consisting of these three true/false questions: i. I am participating in a clinical trial and may be selected to receive the Sanvello app or wait for 8 weeks to receive access to the app. (T) ii. I am a volunteer and can drop out of the study at any time, without penalty. (T) iii. I will be completing questionnaires every 2 weeks and will receive either Amazon gift codes or Visa giftcards as payment for answering questions. (T)
4. Participants who agree to participate will be directed to complete other screening/eligibility questions (uploaded for review)
5. Eligible participants are directed to online baseline assessment

   1. We will collect participant email address for future automated assessment invitations (from REDCap) and for issuing incentive payments for completed assessments.
   2. We will assess further eligibility criteria, including the PHQ-9 and GAD-7 (uploaded for review)
   3. Eligible participants will complete online baseline assessment
   4. Participants (up to 375) will be randomized to one of two groups:
   5. Eligible participants will be randomized according to a computer-generated randomization sequence using randomly permuted blocks, allowing for equal allocation of participants to treatment groups (n = 125 assigned to each treatment group). The randomization sequence will be created by the graduate research assistant using R statistical software. Randomization assignment will be concealed until after entry criteria are confirmed.
   6. Participants in the trial will be randomly assigned to either a) receive the self-guided app intervention immediately, or b) receive the self-guided intervention after an 8-week waiting period (waitlist control group). All groups will have a total of 8 weeks participating in the study, and will complete assessments every 2 weeks during that 8-week period.
   7. Unique study IDs are automatically assigned to each participant at this point. This study ID will link their assessment data and their Sanvello app data.
   8. Participants will receive an electronic invitation (link) to either a) download the self-guided app; or b) notifications of waitlist condition. These invitations will contain unique participant identifiers to link to their Sanvello app data
6. All participants receive biweekly notifications for assessments (weeks 2, 4, 6, and 8). These are sent automatically from REDCap to the email address that the participant provided at baseline.

   a. Participants will have one week to complete the schedule assessment at each timepoint before the assessment window closes.
7. At the end of 8-week study participation, individuals assigned to the waitlist control will receive a promo code for 8 weeks of complimentary Sanvello use. This code will include the unique participant ID, which will be used to track Sanvello app use. This is provided as a benefit of participation. No further data will be collected after the 8-week control condition timeframe ends.
8. The graduate research assistant will send participant incentive (for completed assessment) via email on a biweekly basis based on assessment completion records in REDCap.
9. At the end of study data collection, the PI will destroy the record of participant email addresses as the only identifying link to study records.
10. After data collection has stopped, all incentives have been issued, and the link to the identifier (i.e., email addresses) has been destroyed, Sanvello will send a deidentified dataset to the PI using their secure data transfer system.

    1. This dataset will include unique participant IDs and deidentified usage analytics, including number of app sessions, number of days the intervention was used, time to last use, days of app use, and completion of app tasks. These data are routinely collected from all users per Sanvello's Privacy Policy.

Dr. Renn (PI) and Dr. Raue (Co-I) will meet with the Sanvello team at least twice during data collection to discuss recruitment and study progress. The Sanvello team consists of the company's Chief Medical Officer and Chief Technology Officer, in addition to a project manager and other staff as necessary.

Study Assessments:

For this study, participants will complete a screener to determine potential eligibility, delivered as an online questionnaire., details about their smartphone use, and psychopathology for study eligibility (i.e. a self-report measure of depression (Patient Health Questionnaire (PHQ)-8 score ≥10) and a self-report measure of anxiety (Generalized Anxiety Disorder (GAD) 7-item Scale score ≥8)), in addition to questions about diagnoses and mental health treatment that would render them ineligible.

Following the screener, individuals who are eligible for study participation will be provided the online consent form. Individuals who consent to the study will then be invited to complete the baseline assessment and randomized into the longitudinal trial.

Eligible individuals will be asked to provide their contact (email) and demographic information.

Participants completing the longitudinal study will complete follow-up assessments via online questionnaires at Weeks 2, 4, 6, and 8.

ELIGIBILITY:
Inclusion Criteria:

* • Have a compatible smartphone (Android or Apple)

  * Age 18 or older
  * Ability to read and write English [Justification: (1) limited availability of Sanvello coaches fluent in languages other than English; and (2) use of English language assessments.]
  * Located in the US
  * Clinically significant symptoms of depression and/or anxiety, as evidenced by:

    1. Scores of ≥10 on the PHQ-9 depression assessment (Kroenke et al., 2009); and/or
    2. Scores of ≥8 on the GAD-7 anxiety assessment (Spitzer et al., 2006)

Exclusion Criteria:

* • Active suicidal ideation

  * History of suicide attempt(s)
  * Current symptoms of:

    1. Psychosis
    2. Active substance abuse
  * History of provider diagnosis of:

    1. Bipolar disorder ("manic-depression")
    2. Dementia
    3. Intellectual disability
  * Currently in or scheduled to initiate individual psychotherapy to avoid treatment interference.
  * Prior use of Sanvello
  * Psychotropic medication permitted if dose was stable over the past 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4607 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Depression scores on the Patient Health Questionnaire-9 (PHQ-9) at end of treatment | 8 weeks
  Participants self-reported depression symptoms. Scores range from 0 to 27 where higher scores indicate poorer outcomes (more severe depression).
Anxiety scores from the General Anxiety Disorder-7 (GAD-7) at the end of treatment | 8 weeks
  Participants self-reported anxiety symptoms. Scores range from 0 to 21 where higher scores indicate poorer outcomes (i.e., more severe anxiety).

SECONDARY OUTCOMES:
Health-related quality of life scores from The Patient Reported Outcomes Measurement Information System (PROMIS) Global Health measure at the end of treatment | 8 weeks
  Participants self-reported their global physical, mental, and social health-related quality of life (H-RQoL). Higher T-scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Brenna Renn, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Renn BN, Walker TJ, Edds B, Roots M, Raue PJ. Naturalistic use of a digital mental health intervention for depression and anxiety: A randomized clinical trial. J Affect Disord. 2025 Jan 1;368:429-438. doi: 10.1016/j.jad.2024.09.104. Epub 2024 Sep 17. PMID 39299591